CLINICAL TRIAL: NCT03166761
Title: Randomized Prospective Study of Particulate Corticosteroid Versus Non-particulate Corticosteroid for Sacroiliac Joint Steroid Injection
Brief Title: Particulate Corticosteroid Versus Non-particulate Corticosteroid for Sacroiliac Joint Injection
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment and staffing
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Byron Schneider, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCHNEIBJ03152017153735
Record Dates: First submitted 2017-05-16; First posted 2017-05-25 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Sacro-Iliac Spondylosis
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Experimental): dexamethasone injected into the sacroiliac joint
  Interventions: Drug: Dexamethasone
- Triamcinolone (Active Comparator): triamcinolone injected into the sacroiliac joint
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone injection into the sacroiliac joint
  Other Names: decadron
  Arms: Dexamethasone
Drug: Triamcinolone Acetonide — Triamcinolone injection into the sacroiliac joint
  Other Names: Kenalog
  Arms: Triamcinolone

SUMMARY:
Comparing two different corticosteroids (dexamethasone and triamcinolone) for use in sacroiliac joint injections

DETAILED DESCRIPTION:
Patients eligible for a sacroiliac joint injection will be randomized to receive one of two different steroids, dexamethasone or triamcinolone. The response immediately after injection will be assessed to confirm the diagnosis, and then they will be followed for three month to assess the degree of pain relief experienced

ELIGIBILITY:
Inclusion Criteria:

* Aged >18, capable of understanding and providing consent in English, capable of complying with the outcome instruments used, capable of attending all planned follow up visits
* Unilateral low back/buttocks pain of at least 2 weeks.
* Patient reported 7 day average of numeric pain rating score (NPRS) low back/buttocks pain of at least 5/10 at baseline evaluation
* Clinical diagnosis of sacroiliac joint pain as diagnosed by a board certified Physiatrist including history of low back/buttocks pain and at least 2 positive physical exam findings (including positive fortin finger sign, pain with palpation of posterior superior iliac spine, positive FABER's test, positive Gaenslan's test, positive sacral distraction, positive thigh thrust, positive lateral compression, positive sacral thrust)
* Patient consents to sacroiliac joint corticosteroid injection in a shared decision-making process with the treating physician.
* 80% or more relief of index pain within first 5-15 minutes after injection

Exclusion Criteria:

* Clinical suspicion of alternative process is greater than clinical suspicion of sacroiliac joint pain
* Those receiving remuneration for their pain treatment (e.g., disability, worker's compensation).
* Those involved in active litigation relevant to their pain.
* Those unable to read English and complete the assessment instruments.
* Those unable to attend follow up appointments
* The patient is incarcerated.
* History of prior sacroiliac joint fusion
* Progressive lower extremity neurologic deficit (from active radiculopathy, unhealed radiculopathy, or neuromuscular disease)
* Sacroiliac joint steroid injection within the prior 12 months
* 2 Positive lumbar medial branch blocks within the past 12 months
* Radiofrequency ablation of the lumbar spine within the past 12 months
* Lumbar facet steroid injections within the past 12 months
* Prior epidural steroid injection within the prior 3 months in any location within the spine.
* Possible pregnancy or other reason that precludes the use of fluoroscopy.
* Allergy to steroid, contrast media, or local anesthetics.
* BMI>40.
* Systemic inflammatory arthritis (e.g., rheumatoid arthritis, ankylosing spondylitis, lupus).
* Active infection or treatment of infection with antibiotics within the past 7 days.
* Medical conditions causing significant functional disability (e.g., stroke, decompensated COPD, decompensated heart failure)
* Chronic widespread pain or somatoform disorder (e.g. fibromyalgia).
* Addictive behavior, severe clinical depression, or psychotic features.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Byron Schneider, Principal Investigator — Assistant professor
Locations (1):
- Byron Schneider, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 18 of the 41 patients enrolled had a negative diagnostic response to initial injection and were not followed due to the negative screen after enrollment
Period: Overall Study
Arm/Group | Dexamethasone | Triamcinolone
Started | 9 | 14
Completed | 9 | 10
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Population: the other 18 patients with a negative diagnostic response were not included in the study after the negative screen
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone | Triamcinolone | Total
Number analyzed (Participants) | 9 | 14 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (19.1) | 56.5 (15.7) | 57.8 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 13 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pain Using Numeric Pain Rating Score
Description: Numeric pain rating score, 11 point scale (0-10) filled out on a form indicating the degree of relief/discomfort after the injection. Pain was assessed monthly from baseline to 3 months following the injection. The average value at month 3 is reported.
Time Frame: Baseline to 3 months; Average value at month 3 reported
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexamethasone | Triamcinolone
Number analyzed (Participants) | 9 | 10
units on a scale | 4.2 (2.7) | 4.4 (2.1)

ADVERSE EVENTS:
Time Frame: baseline to 3 months
Arm/Group | Dexamethasone | Triamcinolone
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/14
Other Adverse Events (participants affected / at risk) | 0/9 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT03166761/Prot_SAP_001.pdf